CLINICAL TRIAL: NCT06595433
Title: Effect of Post-Activation Potentiation Effect on Snatch Performance to Exhaustion in Elite Weightlifters
Brief Title: Effect of Post-Activation Potentiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Zarife Pancar, Associate Professor, University of Gaziantep
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: GAUN-SBF-PANCAR-01
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post-Activation Potentiation; Performance
Keywords: Weightlifting, snatch, training

STUDY DESIGN:
Intervention Model Description: The study was designed according to a randomized crossover experimental design. All study sessions were conducted in the fitness center in the weightlifting hall.
Who Masked: Participant
Masking Description: Weightlifters were randomly divided into three groups (A, B, C) of four people. Throughout the study, all groups practiced each warm-up protocol sequentially on different days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PAPE 90% warm up protocol (Experimental): performed three repetitions of dip squats with 90% of their one-repetition maximal dip squats and rested for 4 minutes.
  Interventions: Other: Experimental
- PAPE 50% warm up protocol (Experimental): performed three repetitions of dip squats with 50% of their one-repetition maximal dip squats and rested for 4 minutes.
  Interventions: Other: Experimental
- Unloaded warm-up protocol (Other): They performed the snatch movement with 75% of their maximum snatch weight without pre-warm-up, i.e. without weights, until exhaustion.
  Interventions: Other: unloaded protocol

INTERVENTIONS:
Other: Experimental — In the PAPE 90% protocol, participants performed a general warm-up (e.g., jogging on a treadmill) for 5 minutes and a weightlifting-specific warm-up for 5 minutes, followed by 2 minutes of rest. After resting, they were asked to perform ten repetitions of dip squats with body weight and rested for 1 minute.Then, unlike the unloaded protocol, they performed three repetitions of dip squats with 90% of their one-repetition maximal dip squats and rested for 4 minutes. After resting, they performed a snatch to exhaustion with 75% of their maximum snatch weight. Then they rested for 2 minutes and performed one more repetition of the snatch to exhaustion. The maximum number of repetitions between sets was recorded.
  Arms: PAPE 90% warm up protocol
Other: Experimental — In the PAPE 50% protocol, 5 minutes of general warm-up (jogging on a treadmill) and 5 minutes of weightlifting-specific warm-up were followed by 2 minutes of rest as in the other protocols. After resting, they were asked to perform ten repetitions of body-weighted dip squats and rested for 1 minute. Then, unlike the unloaded and PAPE 90% protocols, they performed eight repetitions of bottom squats with 50% of their maximal bottom squats for one repetition and rested for 4 minutes. After resting, they performed snatches with 75% of their maximum snatch weight until exhaustion. Then they rested for 2 minutes and performed one more repetition of the snatch to exhaustion. The maximum number of repetitions was recorded for statistical analysis.
  Arms: PAPE 50% warm up protocol
Other: unloaded protocol — In the unloaded protocol, subjects performed a 5-minute general warm-up (e.g., jogging on a treadmill) and 5 minutes of weightlifting-specific warm-up followed by 2 minutes of rest. After resting, they performed ten repetitions of bottom squats with their body weight and then rested for 1 minute. After rest, they performed the snatch movement with 75% of their maximum snatch weight until exhaustion. Then, they rested for 2 minutes and again performed the snatch with 75% of their maximum snatch weight until exhaustion. The maximum number of snatch repetitions performed by the weightlifters was recorded for statistical analysis.
  Arms: Unloaded warm-up protocol

SUMMARY:
This study investigated the acute effect of post-activation performance enhancement (PAPE) on snatch performance to exhaustion in elite weightlifters.

DETAILED DESCRIPTION:
Background This study investigated the acute effect of post-activation performance enhancement (PAPE) on snatch performance to exhaustion in elite weightlifters.

Methods The study was designed according to a randomized crossover experimental design. Twelve male elite athletes (age; 18.45 ± 0.52 years; height; 1.73 ± 0.03m, body mass; 71.36 ± 11.36kg) voluntarily participated in the study. The participants performed a general warm-up for five minutes, followed by a weightlifting-specific warm-up for five minutes, and rested for two minutes. Then, the athletes performed three different PAPE protocols on different days and performed the snatch performance to exhaustion. Shapiro-Wilk test was applied for the normality test, and the Levene test was applied for the homogeneity test. Repeated measures of two-way analysis of variance (2x3) were applied to analyze the differences between treatments. Greenhouse-Geiser correction test was used for measurements where the sphericity assumption was not met.

ELIGIBILITY:
Inclusion Criteria:

* no recent injury
* no medication or supplements
* being a volunteer

Exclusion Criteria:

* doping or chronic drug use
* neuromuscular disease, metabolic, hormonal, or cardiovascular disorders,
* and orthopedic limitation

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
number of snatch repetitions performed to exhaustion | Two weeks
  This outcome is measured to determine how different warm-up protocols (90% 1RM squats, 50% 1RM squats, and no-load condition) affect the athletes' performance in snatch repetitions. The statistical analysis focuses on comparing the average number of repetitions between these protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Zarife Pancar, PhD, Study Director — Sports Sciences Research Center
Locations (1):
- Gaziantep University, Faculty of Sport Sciences, Gaziantep, Sehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No